CLINICAL TRIAL: NCT00848276
Title: Human Studies On Gender Differences In PCSK9 Function In Lipoprotein Metabolism
Brief Title: Sex Hormones and Blood PCSK9 Levels
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: T.C. Ooi, Ottawa Hospital Research Institute
Other Study IDs: 2008138-01H
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Hypercholesterolemia
Keywords: PCSK9; Lipoprotein metabolism; testosterone; estradiol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Hypogonadal Men before and after starting testosterone replacement therapy
- 2: Post-menopausal women before and after starting Estrogen Replacement Therapy

SUMMARY:
This study measures a recently discovered protein named PCSK9 (Proprotein convertase subtilisin kexin 9) in blood to see if it is influenced by male and female sex hormones. PCSK9 has recently been shown to control cholesterol and triglyceride levels by diminishing the ability of liver cells to remove cholesterol from blood leading to high blood cholesterol levels.

It was found in previous studies that there was a relationship between blood levels of PCSK9 and cholesterol in men but not in women. This gender difference is a new finding and it raises the question of whether male and female hormones might influence PCSK9's role as a blood cholesterol regulator.

The study requires a pre-treatment fasting blood sample and another sample 3 months after starting hormone therapy.

DETAILED DESCRIPTION:
Proprotein convertase subtilisin kexin 9 (PCSK9) is a secreted glycoprotein that was first demonstrated to play a role in lipoprotein metabolism in 2003 when several gain-of-function single nucleotide polymorphisms (SNPs) in PCSK9 were shown to associate with autosomal dominant hypercholesterolemia (ADH). Soon after, loss-of-function nonsense and missense SNPs in PCSK9 were shown to associate with hypocholesterolemia. Much is still not known about PCSK9's mechanism of action, its substrate(s), its regulation, and factors affecting its function, but we do know that PCSK9 decreases LDL clearance through degradation of LDL receptors. We examined plasma PCSK9 and serum lipids in182 normolipidemic subjects (98 men, 84 women) and found with Spearman analysis a significant correlation between plasma PCSK9 and total cholesterol (TC), LDL-C, and TC/HDL-C in men but not in women, suggesting a gender difference in PCSK9 regulation and/or function.

Following on our unexpected but novel and exciting observation, we hypothesize: that serum levels of testosterone and estradiol would be significantly correlated with plasma PCSK9 levels, that testosterone and 17-B estradiol replacement therapies in men and women respectively would result in changes in the levels of plasma PCSK9, that testosterone and estradiol modify the effect of PCSK9 on serum lipids in different ways, explaining at least in part, the gender dichotomy in PCSK9 function, and that a significant percentage of the effect of hormone replacement therapy on lipids is mediated through PCSK9 function.

Cohort #1 will be 60 hypogonadal men and cohort #2 will be 60 postmenopausal (hypoestrogenic) women before and after testosterone and estrogen replacement therapy respectively. They will undergo measurements of plasma PCSK9, serum testosterone in men or estradiol in women and TC, triglycerides, HDL-C and LDL-C before and 3 months after starting on replacement therapy. These panel studies will allow us to evaluate whether (a) hormone replacement therapy has an effect on PCSK9, and (b) whether resulting changes in PCSK9 are then associated with lipid response.

ELIGIBILITY:
Inclusion Criteria:

Males:

* 18 years of age and older for hypogonadal males/males with prostate cancer
* Prior clinical decision to start on testosterone therapy

Females:

* 30 years of age and older for post-menopausal women
* Prior clinical decision to start on estrogen therapy

Exclusion Criteria:

* Cognitive impairment, active or chronic hepatic or renal disease, diagnosed diabetes mellitus,alcohol consumption greater than 4 drinks/day
* receiving or needing progestogen therapy for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clincs
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teik Chye Ooi, MBBS, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Riverside Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Ooi TC, Raymond A, Cousins M, Favreau C, Taljaard M, Gavin C, Jolly EE, Malone S, Eapen L, Chretien M, Mbikay M, Mayne J. Relationship between testosterone, estradiol and circulating PCSK9: Cross-sectional and interventional studies in humans. Clin Chim Acta. 2015 Jun 15;446:97-104. doi: 10.1016/j.cca.2015.03.036. Epub 2015 Apr 7. PMID 25858546